CLINICAL TRIAL: NCT00824655
Title: A Phase 3, Open-Label Trial, Evaluating the Safety, Tolerability, and Immunogenicity of 13-valent Pneumococcal Conjugate Vaccine in Healthy Children Previously Partially Immunized With Prevenar
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth, Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6096A1-3012
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2011-07-18 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Pneumococcal Vaccines
Keywords: Healthy Subjects; Vaccines; Pneumococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Biological: 13vPnC
- Group 2 (Experimental)
  Interventions: Biological: 13vPnC

INTERVENTIONS:
Biological: 13vPnC — 13vPnC will be administered by intramuscular injection at approximately 5 and 12 months of age.
  Arms: Group 1
Biological: 13vPnC — 13vPnC will be administered by intramuscular injection at approximately 12 months of age.
  Arms: Group 2

SUMMARY:
The purposes of this study are to evaluate the safety of 13-valent pneumococcal Conjugate Vaccine (13vPnC) in children who have already been vaccinated with Prevenar. The study will also assess the immunological response (measure the amount of antibodies, i.e. proteins that fight off germs) produced by children after they have been given the 13-valent pneumococcal vaccine at 5 and 12 months or 12 months of age. In addition, reactions at the injection site will be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children previously immunized with 1 or 2 doses of Prevenar.
* Group 1: Male or female subjects between the age of >=140 and <=196 days of age at time of enrollment.
* Group 2: Male or female subjects between the age of >=336 and <=392 days of age at time of enrollment
* Available for entire study period.

Exclusion Criteria:

* Previous reaction or contra-indication to pneumococcal vaccine or vaccine related component.
* Previous vaccination with licensed or investigational pneumococcal vaccine other than Prevenar.

Ages: 140 Days to 392 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 234 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Sweden (7):
  - Pfizer Investigational Site, Eskilstuna
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Örebro
  - Pfizer Investigational Site, Östersund
  - Pfizer Investigational Site, Uddevalla
  - Pfizer Investigational Site, Umeå

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3012&StudyName=Study%20Evaluating%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20in%20Healthy%20Children

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Group 1 participants received 1 dose of Prevenar at least 42 days prior to study enrollment. Group 2 participants received 2 doses of Prevenar with the last dose at least 140 days prior to study enrollment.
Groups:
- 13vPnC/13vPnC: Participants received two doses of 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) intramuscularly (IM) at 5 months (Infant dose) and 12 months (Toddler dose) of age. Participants had received a single dose of Prevenar, 7-valent pneumococcal conjugate vaccine (7vPnC), at approximately 3 months of age prior to enrollment in the study.
- 13vPnC: Participants received one dose of 13vPnC 0.5 mL IM at 12 months (Toddler dose) of age. Participants had received Prevenar, 7vPnC, at approximately 3 and 5 months of age prior to enrollment in the study.
Period: Infant Series (5 Months of Age)
Arm/Group | 13vPnC/13vPnC | 13vPnC
Started | 118 | 0
Completed | 118 | 0
Not Completed | 0 | 0
Period: After Infant Dose (6 Months of Age)
Arm/Group | 13vPnC/13vPnC | 13vPnC
Started | 118 | 0
Completed | 118 | 0
Not Completed | 0 | 0
Period: Toddler Dose (12 Months of Age)
Arm/Group | 13vPnC/13vPnC | 13vPnC
Started | 118 | 116
Completed | 116 | 116
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Parent/legal guardian request | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 13vPnC/13vPnC: Participants received two doses of 13vPnC 0.5 milliliter (mL) intramuscularly (IM) at 5 months (Infant dose) and 12 months (Toddler dose) of age. Participants had received a single dose of Prevenar, 7vPnC, at approximately 3 months of age prior to enrollment in the study.
- 13vPnC: Participants received one dose of 13vPnC 0.5 mL IM at 12 months (Toddler dose) of age. Participants received Prevenar, 7vPnC, at approximately 3 and 5 months of age prior to enrollment in the study.
- Total: Total of all reporting groups
Arm/Group | 13vPnC/13vPnC | 13vPnC | Total
Number analyzed (Participants) | 118 | 116 | 234
Age Continuous [Mean (Standard Deviation); unit: months] | 5.1 (0.37) | 11.9 (0.52) | 8.5 (3.42)
Sex/Gender, Customized [Number; unit: participants]
  Female | 50 | 60 | 110
  Male | 68 | 56 | 124

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-Specific Pneumococcal Immunoglobulin G (IgG) Antibodies 1 Month After the Toddler Dose
Description: Antibody geometric mean concentration (GMC) as measured by micrograms per milliliter (mcg/mL) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) were presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. GMCs were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: Evaluable Toddler Immunogenicity Population: eligible participants who received study vaccine at the expected dose(s), blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC/13vPnC | 13vPnC
Number analyzed (Participants) | 114 | 115
mcg/mL
  Common Serotype 4 | 5.27 [4.43 to 6.26] | 5.06 [4.22 to 6.06]
  Common Serotype 6B | 9.63 [8.01 to 11.57] | 8.75 [6.76 to 11.32]
  Common Serotype 9V | 3.50 [3.01 to 4.07] | 3.33 [2.88 to 3.84]
  Common Serotype 14 | 9.22 [7.66 to 11.09] | 9.30 [7.90 to 10.95]
  Common Serotype 18C | 2.93 [2.50 to 3.44] | 3.87 [3.30 to 4.53]
  Common Serotype 19F | 7.70 [6.12 to 9.69] | 8.31 [6.39 to 10.81]
  Common Serotype 23F | 3.27 [2.68 to 3.99] | 4.40 [3.70 to 5.22]
  Additional Serotype 1 | 14.65 [12.50 to 17.17] | 1.58 [1.30 to 1.93]
  Additional Serotype 3 | 1.85 [1.59 to 2.15] | 1.34 [1.13 to 1.58]
  Additional Serotype 5 | 7.02 [5.98 to 8.25] | 1.44 [1.21 to 1.72]
  Additional Serotype 6A | 6.14 [5.08 to 7.43] | 2.48 [1.89 to 3.26]
  Additional Serotype 7F | 5.86 [5.11 to 6.72] | 3.55 [3.09 to 4.08]
  Additional Serotype 19A | 7.25 [6.14 to 8.57] | 13.16 [11.26 to 15.38]

2. Secondary Outcome: Percentage of Participants Achieving a Serotype-specific IgG Antibody Greater Than or Equal To (≥) 0.35 Mcg/mL, 1 Month After the Infant Dose
Description: Percentage of participants achieving predefined antibody threshold ≥0.35 mcg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: 1 Month after the infant series (6 months of age)
Population: Evaluable Infant Immunogenicity Population: eligible participants who received study vaccine at the expected dose(s), blood drawn within specified timeframes, at least 1 valid and determinate assay result for proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC/13vPnC
Number analyzed (Participants) | 115
Percentage of participants
  Common Serotype 4 | 99.1 [95.3 to 100.0]
  Common Serotype 6B | 53.0 [43.5 to 62.4]
  Common Serotype 9V | 99.1 [95.3 to 100.0]
  Common Serotype 14 | 96.5 [91.3 to 99.0]
  Common Serotype 18C | 95.7 [90.1 to 98.6]
  Common Serotype 19F | 92.2 [85.7 to 96.4]
  Common Serotype 23F | 62.6 [53.1 to 71.5]
  Additional Serotype 1 | 80.9 [72.5 to 87.6]
  Additional Serotype 3 | 100.0 [96.8 to 100.0]
  Additional Serotype 5 | 83.5 [75.4 to 89.7]
  Additional Serotype 6A | 36.8 [28.0 to 46.4]
  Additional Serotype 7F | 93.0 [86.8 to 96.9]
  Additional Serotype 19A | 87.8 [80.4 to 93.2]

3. Secondary Outcome: GMC of Serotype-Specific Pneumococcal IgG Antibodies Measured 1 Month After the Infant Dose
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) presented. GMC (13vPnC) and corresponding 2-sided 95% confidence intervals (CI) were evaluated. GMCs calculated using all participants with available data for the specified blood draw.
Time Frame: 1 Month after the infant series (6 months of age)
Population: Evaluable Infant Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC/13vPnC
Number analyzed (Participants) | 115
mcg/mL
  Common Serotype 4 | 2.90 [2.48 to 3.40]
  Common Serotype 6B | 0.40 [0.32 to 0.50]
  Common Serotype 9V | 1.73 [1.50 to 1.99]
  Common Serotype 14 | 4.70 [3.72 to 5.92]
  Common Serotype 18C | 1.56 [1.29 to 1.89]
  Common Serotype 19F | 3.01 [2.34 to 3.88]
  Common Serotype 23F | 0.57 [0.46 to 0.70]
  Additional Serotype 1 | 0.89 [0.73 to 1.08]
  Additional Serotype 3 | 1.88 [1.65 to 2.14]
  Additional Serotype 5 | 0.72 [0.62 to 0.84]
  Additional Serotype 6A | 0.28 [0.23 to 0.34]
  Additional Serotype 7F | 1.78 [1.48 to 2.15]
  Additional Serotype 19A | 0.85 [0.73 to 0.99]

4. Secondary Outcome: GMC of Serotype-Specific Pneumococcal IgG Antibodies Measured Before the Toddler Dose
Description: Antibody GMC for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) presented. GMC (13vPnC) and corresponding 2-sided 95% CIs evaluated. GMCs calculated using all participants with available data for the specified blood draw.
Time Frame: 12 months of age (prior to toddler dose)
Population: Evaluable Toddler Immunogenicity Population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC/13vPnC | 13vPnC
Number analyzed (Participants) | 114 | 115
mcg/mL
  Common Serotype 4 | 0.66 [0.57 to 0.77] | 0.62 [0.53 to 0.72]
  Common Serotype 6B | 0.83 [0.67 to 1.02] | 0.65 [0.51 to 0.82]
  Common Serotype 9V | 0.74 [0.65 to 0.85] | 0.70 [0.60 to 0.82]
  Common Serotype 14 | 1.99 [1.63 to 2.42] | 2.23 [1.85 to 2.69]
  Common Serotype 18C | 0.35 [0.30 to 0.41] | 0.44 [0.38 to 0.51]
  Common Serotype 19F | 0.85 [0.70 to 1.03] | 0.81 [0.66 to 1.00]
  Common Serotype 23F | 0.33 [0.27 to 0.39] | 0.41 [0.34 to 0.49]
  Additional Serotype 1 | 0.46 [0.40 to 0.53] | 0.01 [0.01 to 0.02]
  Additional Serotype 3 | 0.40 [0.34 to 0.47] | 0.05 [0.04 to 0.07]
  Additional Serotype 5 | 1.18 [1.02 to 1.36] | 0.33 [0.26 to 0.42]
  Additional Serotype 6A | 0.71 [0.60 to 0.85] | 0.24 [0.19 to 0.31]
  Additional Serotype 7F | 1.08 [0.95 to 1.23] | 0.02 [0.02 to 0.02]
  Additional Serotype 19A | 1.06 [0.88 to 1.28] | 1.55 [1.32 to 1.81]

5. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions: Infant Series Dose 1 (5 Months of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may have been represented in more than 1 category.
Time Frame: Day 1 through Day 7 after vaccination
Population: Safety Population: all participants who received at least 1 dose of the study vaccine; n = number of participants reporting yes for at least 1 day or no for all days for the specific characteristic
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC/13vPnC
Number analyzed (Participants) | 113
Percentage of participants
  Tenderness: Any (n=108) | 36.1
  Tenderness: Significant (n=99) | 3.0
  Swelling: Any (n=104) | 33.7
  Swelling: Mild (n=104) | 31.7
  Swelling: Moderate (n=101) | 9.9
  Swelling: Severe (n=99) | 0.0
  Redness: Any (n=107) | 40.2
  Redness: Mild (n=107) | 36.4
  Redness: Moderate (n=99) | 4.0
  Redness: Severe (n=99) | 0.0

6. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 7 Days of the Toddler Dose (12 Months of Age)
Description: as for outcome 5
Time Frame: Day 1 through Day 7 after vaccination
Population: Safety Population; n = number of participants reporting yes for at least 1 day or no for all days for the specific characteristic
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC/13vPnC | 13vPnC
Number analyzed (Participants) | 108 | 115
Percentage of participants
  Tenderness: Any (n=104,110) | 59.6 | 52.7
  Tenderness: Significant (n=96,103) | 5.2 | 7.8
  Swelling: Any (n=104,110) | 53.8 | 54.5
  Swelling: Mild (n=104,109) | 50.0 | 52.3
  Swelling: Moderate (n=100,105) | 24.0 | 29.5
  Swelling: Severe (n=95,101) | 0.0 | 0.0
  Redness: Any (n=104,113) | 62.5 | 59.3
  Redness: Mild (n=103,113) | 52.4 | 51.3
  Redness: Moderate (n=98,106) | 20.4 | 26.4
  Redness: Severe (n=95,101) | 0.0 | 0.0

7. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 7 Days of the Infant Dose (5 Months of Age)
Description: Systemic events (any fever ≥ 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, and decreased sleep) were reported using an electronic diary. Participants may have been represented in more than 1 category.
Time Frame: Day 1 through 7 after vaccination
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC/13vPnC
Number analyzed (Participants) | 117
Percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C (n=103) | 26.2
  Fever >39 degrees C but ≤40 degrees C (n=99) | 2.0
  Fever >40 degrees C (n=99) | 0.0
  Decreased appetite (n=107) | 36.4
  Irritability (n=114) | 80.7
  Increased sleep (n=106) | 50.9
  Decreased sleep (n=112) | 39.3

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 7 Days of the Toddler Dose (12 Months of Age)
Description: Systemic events (any fever ≥ 38 degrees C, decreased appetite, irritability, increased sleep, and decreased sleep) were reported using an electronic diary. Participants may have been represented in more than 1 category.
Time Frame: Day 1 through 7 after vaccination
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC/13vPnC | 13vPnC
Number analyzed (Participants) | 113 | 114
Percentage of participants
  Fever ≥38 degrees C but ≤39 degrees C (n=99,105) | 31.3 | 32.4
  Fever >39 degrees C but ≤40 degrees C (n=96,102) | 5.2 | 3.9
  Fever >40 degrees C (n=95,101) | 0.0 | 0.0
  Decreased appetite (n=103,109) | 46.6 | 44.0
  Irritability (n=111,113) | 82.0 | 76.1
  Increased sleep (n=101,108) | 49.5 | 38.9
  Decreased sleep (n=105,106) | 36.2 | 33.0

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- 13vPnC/13vPnC at 5 Months: 13vPnC 0.5 mL dose administered IM at 5 months of age (infant dose)
- 13vPnC/13vPnC at 6 Months of Age: 13vPnC 0.5 mL dose administered IM at 5 months of age (infant dose); assessment 1 month after the infant series (6 months of age).
- 13vPnC/13vPnC at 12 Months: 13vPnC 0.5 mL dose administered IM at 5 months (infant dose) and 12 months of age (toddler dose).
- 13vPnC at 12 Months: 13vPnC 0.5 mL dose administered IM at 12 months of age (toddler dose).
Arm/Group | 13vPnC/13vPnC at 5 Months | 13vPnC/13vPnC at 6 Months of Age | 13vPnC/13vPnC at 12 Months | 13vPnC at 12 Months
Serious Adverse Events (participants affected / at risk) | 1/118 | 4/118 | 1/116 | 0/116
Other Adverse Events (participants affected / at risk) | 92/118 | 4/118 | 91/116 | 86/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC/13vPnC at 5 Months (N=118) | 13vPnC/13vPnC at 6 Months of Age (N=118) | 13vPnC/13vPnC at 12 Months (N=116) | 13vPnC at 12 Months (N=116)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 4 | 0 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC/13vPnC at 5 Months (N=118) | 13vPnC/13vPnC at 6 Months of Age (N=118) | 13vPnC/13vPnC at 12 Months (N=116) | 13vPnC at 12 Months (N=116)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 5 | 0
Pyrexia (General disorders) | 1 | 0 | 4 | 4
Nasopharyngitis (Infections and infestations) | 5 | 0 | 8 | 7
Exanthema subitum (Infections and infestations) | 1 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Crying (Nervous system disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 2 | 3
Otitis media (Infections and infestations) | 0 | 0 | 2 | 2
Varicella (Infections and infestations) | 0 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 39/108 | 0/0 | 62/104 | 58/110
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 3/99 | 0/0 | 5/96 | 8/103
Swelling (Any) (Skin and subcutaneous tissue disorders) | 35/104 | 0/0 | 56/104 | 60/110
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 33/104 | 0/0 | 52/104 | 57/109
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 10/101 | 0/0 | 24/100 | 31/105
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 0/99 | 0/0 | 0/95 | 0/101
Redness (Any) (Skin and subcutaneous tissue disorders) | 43/107 | 0/0 | 65/104 | 67/113
Redness (Mild) (Skin and subcutaneous tissue disorders) | 39/107 | 0/0 | 54/103 | 58/113
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 4/99 | 0/0 | 20/98 | 28/106
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/99 | 0/0 | 0/95 | 0/101
Fever ≥38°C but ≤39°C (General disorders) | 27/103 | 0/0 | 31/99 | 34/105
Fever >39°C but ≤40°C (General disorders) | 2/99 | 0/0 | 5/96 | 4/102
Fever >40°C (General disorders) | 0/99 | 0/0 | 0/95 | 0/101
Decreased appetite (General disorders) | 39/107 | 0/0 | 48/103 | 48/109
Irritability (General disorders) | 92/114 | 0/0 | 91/111 | 86/113
Increased sleep (General disorders) | 54/106 | 0/0 | 50/101 | 42/108
Decreased sleep (General disorders) | 44/112 | 0/0 | 38/105 | 35/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.